CLINICAL TRIAL: NCT01991509
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel Group Study Assessing the Safety, Tolerability and Pharmacokinetics of Two Different Doses of LBR-101 Given Intravenously and Subcutaneously
Brief Title: Safety and Bioavailability of IV and SC LBR-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: LBR-101-011
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Bioavailability and Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- LBR-101 IV Dose 1 (Experimental): LBR-101 Dose 1 Administered Intravenously
  Interventions: Biological: LBR-101 IV
- LBR-101 SC Dose 1 (Experimental): LBR-101 Dose 1 Administered Subcutaneously
  Interventions: Biological: LBR-101 SC
- Placebo IV (Placebo Comparator): Placebo Administered Intravenously
  Interventions: Biological: LBR-101 IV
- Placebo SC (Placebo Comparator): Placebo Administered Subcutaneously
  Interventions: Biological: LBR-101 SC
- LBR-101 Dose 2 IV (Experimental): LBR-101 Dose 2 Administered Intravenously
  Interventions: Biological: LBR-101 IV
- LBR-101 Dose 2 SC (Experimental): LBR-101 Dose 2 Administered Subcutaneously
  Interventions: Biological: LBR-101 SC

INTERVENTIONS:
Biological: LBR-101 IV — LBR-101 Administered Intravenously
  Arms: LBR-101 Dose 2 IV; LBR-101 IV Dose 1; Placebo IV
Biological: LBR-101 SC — LBR-101 Administered Subcutaneously
  Arms: LBR-101 Dose 2 SC; LBR-101 SC Dose 1; Placebo SC

SUMMARY:
The purpose of this study is to assess the safety, tolerability and blood levels of LBR-101 when administered intravenously or subcutaneously to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Generally Healthy, Signed Approved Informed Consent, BMI 17.5-34.5 kg/m2, Willing and able to comply with CRU rules regulations and study schedule

Exclusion Criteria:

* Clinically significant medical or psychiatric condition, Febrile illness within 5 days of dosing, Pregnant or Nursing Females. History of alcoholism, drug addiction or positive drug/alcohol screen, History of hypersensitivity to injected proteins or monoclonal antibodies, Unwilling or unable to comply with the protocol specified lifestyle guidelines, Investigational site staff members, Use of 3 or more prescription or non-prescription medications daily, Acetaminophen use in doses of higher than 1 g or more/day, Daily Aspirin use in higher than 325 mg/day, Treatment with an investigational drug within 30 days of dosing, Use of biologics within 6 months of screening, Any clinically significant abnormality in the 12-Lead ECG, Positive result for HIV, Hepatitis B, or Hepatitis C, Any clinically significant abnormalities in Blood Chemistry Hematology or Urinalysis, Positive Pregnancy Test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of IV versus SC Administration of LBR-101 | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Bigal, MD, PhD, Study Chair — Sponsor Chief Medical Officer; Rafael Escandon, PhD MPH, Study Director — Sponsor Clinical VP
Locations (1):
- PPD Development, Austin, Texas, United States